CLINICAL TRIAL: NCT00160212
Title: A Randomized, Placebo-Controlled, Double-Blind, Six-Arm, Dose Escalation, Multi-Center Study to Evaluate the Efficacy and Safety of SLV306: 150, 300, 600 mg Once Daily, 150-300 mg Twice Daily and Amlodipine 5-10 mg Once Daily in Subjects With Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of SLV306 in Subjects With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S306.2.008; 2004-000305-21
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension
Keywords: blood pressure
MeSH Terms: conditions — Hypertension | interventions — SLV 306

INTERVENTIONS:
Drug: Daglutril

SUMMARY:
This study is to compare the efficacy and safety of increasing doses of SLV306 with amlodipine.

ELIGIBILITY:
Inclusion Criteria:

* sitting office diastolic blood pressure between 90 and 109 mmHg
* office systolic blood pressure between 140 and 179 mmHg
* mean day-time diastolic 24-h ABPM blood pressure >= 85 mmHg inclusive at baseline

Exclusion Criteria:

* known secondary hypertension
* decompensated congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (130):
- Australia (6):
  - Site 705, Bracken Ridge
  - Site 706, Caboolture
  - Site 700, Inala
  - Site 701, Kippa-Ring
  - Site 702, Melbourne
  - Site 703, Nedlands
- Bulgaria (8):
  - Site 952, Haskovo
  - Site 955, Pleven
  - Site 951, Plovdiv
  - Site 956, Plovdiv
  - Site 950, Sofia
  - Site 953, Sofia
  - Site 954, Sofia
  - Site 957, Sofia
- Denmark (3):
  - Site 402, Aalborg
  - Site 401, Ballerup Municipality
  - Site 403, Vejle
- Site 850, Tallinn, Estonia
- Germany (19):
  - Site 119, Aschaffenburg
  - Site 101, Bad Nauheim
  - Site 104, Bad Wörishofen
  - Site 106, Beckum
  - Site 110, Deidesheim
  - Site 107, Karlsruhe
  - Site 118, Kassel
  - Site 109, Krombach
  - Site 113, Ladenburg
  - Site 102, Leipzig
  - Site 112, Lollar
  - Site 114, Magdeburg
  - Site 111, Marburg
  - Site 105, Münster
  - Site 115, Niederstetten
  - Site 120, Rodgau Dudenhofen
  - Site 116, Vellmar
  - Site 103, Wiesbaden
  - Site 117, Wolmirstedt
- Hungary (6):
  - Site 800, Budapest
  - Site 805, Budapest
  - Site 803, Gyöngyös
  - Site 801, Kecskemét
  - Site 804, Pécs
  - Site 802, Székesfehérvár
- Israel (11):
  - Site 300, Ashkelon
  - Site 306, Ashkelon
  - Site 304, Beersheba
  - Site 311, Haifa
  - Site 305, Jerusalem
  - Site 310, Kfar Saba
  - Site 303, Kiryat Ata
  - Site 308, Petah Tikva
  - Site 302, Tel Aviv
  - Site 301, Tel Litwinsky
  - Site 309, Tiberias
- Latvia (6):
  - Site 932, Daugavpils
  - Site 930, Kuldīga
  - Site 931, Riga
  - Site 933, Riga
  - Site 934, Riga
  - Site 935, Riga
- Lithuania (3):
  - Site 920, Kaunas
  - Site 923, Klaipėda
  - Site 921, Vilnius
- Slovakia (8):
  - Site 600, Bratislava
  - Site 601, Bratislava
  - Site 607, Košice
  - Site 608, Košice
  - Site 602, Levice
  - Site 605, Lučenec
  - Site 603, Nové Zámky
  - Site 606, Vráble
- United Kingdom (59):
  - Site 262, Addlestone
  - Site 229, Airdrie
  - Site 234, Alexandria
  - Site 245, Bangor
  - Site 241, Barrhead
  - Site 224, Bath
  - Site 240, Bath
  - Site 230, Bellshill
  - Site 243, Bexhill-on-Sea
  - Site 261, Bexhill-on-Sea
  - Site 255, Blackpool
  - Site 222, Blantyre
  - Site 232, Calderbank
  - Site 236, Chesterfield
  - Site 219, Chippenham
  - Site 256, Chippenham
  - Site 237, Co Tyrone
  - Site 216, Coatbridge
  - Site 238, Cornwall
  - Site 207, Coventry
  - Site 247, Cumbernauld
  - Site 208, Dumbarton
  - Site 235, East Horsley
  - Site 220, Ely
  - Site 257, Frome
  - Site 210, Glasgow
  - Site 221, Glasgow
  - Site 227, Glasgow
  - Site 233, Glasgow
  - Site 251, Glasgow
  - Site 201, Greenisland
  - Site 252, Helensburgh
  - Site 249, Hook
  - Site 226, Maidenhead
  - Site 246, Maidenhead
  - Site 213, Manchester
  - Site 244, Melksham
  - Site 259, Middlesex
  - Site 202, Motherwell
  - Site 206, Motherwell
  - Site 217, Motherwell
  - Site 239, Motherwell
  - Site 231, Paisley
  - Site 250, Paisley
  - Site 242, Penzance
  - Site 218, Plymouth
  - Site 223, Plymouth
  - Site 254, Reading
  - Site 212, Riddrie
  - Site 200, Royal Leamington Spa
  - Site 253, Sandy
  - Site 258, Sheffield
  - Site 205, Slough
  - Site 215, St Just
  - Site 211, Strathaven
  - Site 225, Swansea
  - Site 209, Thornhill
  - Site 248, Woking
  - Site 228, Wokingham